CLINICAL TRIAL: NCT03385356
Title: Impact of Vitamin D Supplementation in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Collaborators: Medical Faculty Maribor (Unknown)
Responsible Party: Principal Investigator, Saša Gselman, M.D., M.D., University Medical Centre Maribor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38602SUN17
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Vitamin D Deficiency
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: 1000 IU/day of Vitamin D vs 4000 IU of Vitamin D /day; IU (international units)
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1000 IU of vitamin D per day (Active Comparator): Half of randomized patients will receive 1000 IU of vitamin D per day
  Interventions: Drug: Vitamin D
- 4000 IU of vitamin D per day (Active Comparator): Half of randomized patients will receive 4000 IU of vitamin D per day
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D supplementation of 1000IU vs 4000IU vitamin D per day for four months during winter time, when levels of vitamin D in serum of MS patients are especially low.
  Other Names: Oleovit D3

SUMMARY:
Vitamin D is important risk factor for developing multiple sclerosis (MS) and for disease progression. Patients with MS who had lower vitamin D levels were at increased risk for more clinical attacks and faster disease progression. It was also shown that patients with MS had lower vitamin D levels in serum than healthy controls. It is not clearly defined, which are the levels of vitamin D in serum, that are high enough to trigger immunomodulatory effect and are safe for patients.

This double-blind randomized clinical trial was designed to compare impact of vitamin D supplementation in two different doses (1000 IU/day vs 4000 IU/day) in patients with relapsing remitting MS. The main goal of this trial is to compare dose response on vitamin D supplementation and to estimate more closely appropriate level of vitamin D in serum which triggers some of experimentally shown immunomodulatory actions.

DETAILED DESCRIPTION:
Vitamin D is important risk factor for developing multiple sclerosis (MS) and for disease progression. Patients with MS who had lower vitamin D levels were at increased risk for more clinical attacks and faster disease progression. It was also shown that patients with MS had lower vitamin D levels in serum than healthy controls. It is not clearly defined, which are the levels of vitamin D in serum, that are high enough to trigger immunomodulatory effect and are safe for patients.

This double-blind randomized clinical trial was designed to compare impact of vitamin D supplementation during four months in winter time in two different doses (1000 IU/day vs 4000 IU/day) in patients with relapsing remitting MS. The main goal of this trial is to compare dose response on vitamin D supplementation and estimate more closely appropriate level of vitamin D in serum which triggers some of experimentally shown immunomodulatory actions. To define immunomodulatory response different laboratory, clinical and genetic tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting MS
* Treatment with immunomodulatory drug
* Age 18-60 years and
* EDSS (Expanded Disability Status Scale) score less than 5.

Exclusion Criteria:

* Use of vitamin D supplements in the past 3 months
* Pregnancy, planning pregnancy or nursing
* Relapse of disease and corticosteroids use in past month
* Active inflammation at the start of the study (flu, cystitis etc.)
* Renal disease
* Elevated levels of calcium or parathormone
* Hypersensitivity to vitamin D preparations
* Switching of immunomodulatory drug in past 3 months
* Other autoimmune disease
* History of hyperparathyroidism, liver disease, tuberculosis, sarcoidosis or kidney stones

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Vitamin D supplementation dose response | 4 months
  Change in vitamin D level in serum after supplementation with 1000IU/day or 4000 IU/day.

CONTACTS AND LOCATIONS:
Overall Officials: Saša Gselman, MD, Principal Investigator — University Medical Centre Maribor
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia